CLINICAL TRIAL: NCT07386613
Title: Investigating the Feasibility of Home Monitoring of Visual Function in Populations at High Risk of Developing Diabetic Retinopathy (DR) Using Novel Game-based Technology (OKKO Health)
Brief Title: Feasibility of Home Monitoring of Visual Function in DR
Status: Completed | Type: Observational
Sponsor: Queen's University, Belfast (Other)
Collaborators: OKKO Health (Industry)
Responsible Party: Principal Investigator, Ruth Hogg, Professor Ruth Esther Hogg, Queen's University, Belfast
Other Study IDs: 307008
Record Dates: First submitted 2026-01-16; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Diabetes (DM); Diabetes Complication; Diabetes (Insulin-requiring, Type 1 or Type 2); Diabetic Retinopathy (DR); Diabetes Pregnancy; Gestational Diabetes Mellitus in Pregnancy; Dialysis Patients
Keywords: Remote monitoring; Digital Health; Visual function; High risk patients; Diabetic retinopathy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Complications; Diabetic Retinopathy; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with diabetes at high risk of retinopathy
  Interventions: Device: Okko Health App

INTERVENTIONS:
Device: Okko Health App — Okko Health digital health app used to assess visual acuity and contrast sensitivity using a mobile phone.

SUMMARY:
Diabetes is a serious condition where patients can develop complications in their body including their eyes which can lead to sight loss. Patients with diabetes are encouraged to attend yearly screening appointments at which signs of Diabetic Retinopathy (DR) are assessed. Attendance at these appointments and at any follow-up appointments can be time-consuming and inconvenient for those working. Better ways to monitor changes in vision are needed. Therefore, we are hoping to develop a set of eye tests that a person with diabetes can complete at home on a smartphone in collaboration with researchers at OKKO Health.

ELIGIBILITY:
Inclusion Criteria:

Study 1:

* The 55 participants with Type 1 or Type 2 diabetes must also be a gestational, or dialysis DR patient.
* Aged 18-70.
* All participants should have access to one of the following devices on a daily basis: iPhone (X, XS, XR, 11, 11 Pro, 11 Pro Max, SE 2020, 12, 12 Pro, 12 Pro Max, 12 mini); iPad (Pro 11-inch 2nd generation, Pro 12.9-inch 4th generation); Samsung Galaxy S8, S9, S10, A20e or A40; Samsung Galaxy Tab S3; Honor 10 Lite; Motorola G6 or G7 Power or Pixel 3a.
* All participants should also have the ability to read and understand in English and be able to give informed consent.
* All participants should also be able to tap the screen of a digital device.
* All gestational and dialysis participants should be willing to undergo handheld retinal imaging, no pupil dilation is required.
* Be willing to use the app from home for up to 6 months in between the participant's regular clinic visits.

Study 2:

* The 35 participants with type 1 or type 2 diabetes should have R0 no retinopathy or R1 background changes (this is stated on the letter they receive from the Diabetic Retinal Screening service).
* Participants must already have a diabetic screening letter dated within 3 months and use a continuous glucose monitor and be willing to share the data from their monitor with the study team. They must also be willing to allow the research team access to their most recent OCT scans which will be accessed by Prof Tunde Peto.
* All participants should have access to one of the following devices on a daily basis: iPhone (X, XS, XR, 11, 11 Pro, 11 Pro Max, SE 2020, 12, 12 Pro, 12 Pro Max, 12 mini); iPad (Pro 11-inch 2nd generation, Pro 12.9-inch 4th generation); Samsung Galaxy S8, S9, S10, A20e or A40; Samsung Galaxy Tab S3; Honor 10 Lite; Motorola G6 or G7 Power or Pixel 3a.
* All participants should also have the ability to read and understand in English and be able to give informed consent.
* All participants should also be able to tap the screen of a digital device

Exclusion Criteria: Study 1 and 2:

* The presence of another ocular disease that impacts vision such as age-related macular degeneration, glaucoma, or active uveitis.
* Participants who are unable to tap a screen.
* Serious life-threatening conditions that would preclude attendance in the longitudinal part of the study.
* Neurological conditions that can impair vision
* Any physical limitation that would make the participant unable to attend clinic visits (e.g., patients with arthritis or neck problems who may be unable to sit for a prolonged period of time).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with type 1 or type 2 diabetes with either no diabetic retinopathy (R0) or early background changes (R1)
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2023-09-09 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Primary Outcome : Explore the feasibility of longitudinal monitoring in hard-to-reach clinical populations by analysing recruitment and retention data, frequency of testing, and factors influencing play frequency and sustained engagement with the app. | 6 months
  Assessment of feasibility
  Feasibility was assessed using recruitment, retention and engagement data from the Dialysis, Pregnancy and CGM high risk groups. Attrition rates from verbal agreement to signed consent and study completion were documented and reasons for dropout were captured through research team notes, participant self-report and follow-up communication.
  Engagement was quantified as the number of OKKO Health app plays over 6 months for each eye in the OKKO Circles Acuity (LogMAR) and the OKKO Contrast Sensitivity (LogCS) games. Participants were requested to play both games at least once a week. The app automatically logged usage data, including total plays and plays per eye.

SECONDARY OUTCOMES:
Secondary Outcome: Explore the acceptability of longitudinal monitoring in populations at risk of DR that are hard to reach through qualitative and interview data. | 6 months
  This study utilized both quantitative and qualitative data to assess acceptability and adherence including The Adherence and Acceptability Questionnaire (AAQ) (adapted from Venkatesh et al., 2003) and The Ease of Use and Acceptability Questionnaire (EUAQ) (modified from Tay et al., 2004).
  The adapted 16-item AAQ asked participants questions about their experience regarding five dimensions or aspects of the app: perceived usefulness, perceived ease of use, adherence, behavioural intention and digital system accessibility. For example, the AAQ questionnaire began with the following statement: "I think that using digital health interventions to monitor my vision weekly could be a good thing". Participants then rated this statement in relation to their experience of using the OKKO Health app on a five-point Likert scale, ranging from 1: 'Strongly Disagree' to '5: 'Strongly Agree'.

OTHER OUTCOMES:
3. Third Outcome Measure: Describe the challenges associated with implementing longitudinal home-based monitoring in high-risk populations, identifying key logistical, behavioural, and technological barriers to engagement. | 6 months
  Given the study's exploratory nature and the lack of suitably developed instruments, open-ended survey questions were added to the adapted EUAQ (Tay et al. 2004). These were administered to capture patients' experiences and potential challenges using the OKKO Health app. They began with the question, 'Did you find the tests easy to do? If no- How?'. This question was followed by a list of seven items such as: 'Did you find any of the tests particularly difficult?'; 'Which was your favourite test? Why?'; 'If you knew you had to continue to carry out these tests for a longer period of time would you be willing to continue?'. A multi-line text entry field was implemented in Qualtrics, which allowed participants responses up to five lines. An analysis of the answers to these questions aided the exploration of challenges to. Implementation. In addition to the open-ended questionnaire responses, supplementary qualitative feedback was recorded using multiple sources, through entries in the r

CONTACTS AND LOCATIONS:
Overall Officials: Professor Ruth E Hogg, PhD, Principal Investigator — Queen's University, Belfast
Locations (3):
- United Kingdom (3):
  - Belfast Health and Social Care Trust, Belfast City Hospital, Belfast, Belfast City
  - Northern Health and Social Care Trust, Antrim Hospital, Antrim, County Antrim
  - Southern Health and Social Care Trust, Craigavon Hospital, Craigavon, County Armagh

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make the individual participant data available as the research is currently being submitted as part of a PhD thesis. The full thesis will be available via open access on the Queen's University Belfast repository.